CLINICAL TRIAL: NCT04494607
Title: Evaluation of the Glycemic Index of Various Types of Pasta in Healthy Volunteers
Brief Title: Glycemic Index of Various Types of Pasta in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Maria Gabriella Caruso, M.D, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC2020_IRCCS
Record Dates: First submitted 2020-06-15; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Glycemic Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test arm (Experimental): Determination of Glycemic and Insulinemic curves under different alimentary intake
  Interventions: Dietary Supplement: lowest Glycemic Index for a selected type fo cereal product

INTERVENTIONS:
Dietary Supplement: lowest Glycemic Index for a selected type fo cereal product — determination of lowest Glycemic Index for a selected type fo cereal product

SUMMARY:
he project aims to evaluate the glycemic index of different types of pasta with different formats and with different types of flour. In particular, we want to know the effect of the format and the different type of flour on the glycemic and insulinemic response.

Specific objective 1: determination of the glycemic index of the product concerned.

Specific objective 2: determination of the insulinemic index of the product concerned.

Specific objective 3: determination of the pasta format and the type of flour with a lower glycemic and insulinemic index.

DETAILED DESCRIPTION:
The study is divided into the following phases:

Phase 1: screening of subjects aimed at identifying possession of the inclusion criteria necessary for participation in the study;

Phase 2: Enrollment of the subject and for each of the enlisted subjects, execution of the first and second determination of the glycemic and insulinemic response curve with the standard glucose solution 30 days apart; 15 days after the second determination of the glycemic and insulinemic response to the glucose load, the assumption of the food test will be performed on which to measure the glycemic index (type of pasta) and evaluation of the glycemic and insulinemic response curve to this food ; finally, after a further 30 days, the third determination of the glycemic and insulinemic response curve will be performed with the standard glucose solution;

Phase 3: statistical processing of the results of phase 2 and determination of the glycemic index and insulinemic index for each type of pasta tested;

Phase 4: description of the results of phase 3 with indication to the supplier company of the pasta format and the type of flour with lower glycemic and insulinemic index.

More phases detailed:

Phase 1 Voluntarily enrolled subjects undergo a clinical history to exclude the pathologies present in the exclusion criteria and a routine blood sample to exclude metabolic alterations affecting the metabolism of sugars, lipids, uric acid, and liver.

Phase 2: The subjects considered suitable to enter the study will be subjected to the administration of the standard glucose solution for the determination of the first glycemic and insulinemic curve. The standard solution consists of 50 g of glucose dissolved in 200 cc of trace mineral water, which the subject will be invited to drink in about 10 minutes. Venous blood samples for the determination of glucose and insulin will be collected at time 0, and then at 15, 30, 45, 60, 90 and 120 minutes from the start of the standard intake of the glucose solution. In case of a normal response to the first determination of the glycemic and insulinemic curve, the subject will continue in the study; otherwise it will be excluded and will be directed to clinical study paths to assess the presence of any pathologies not yet concluded (diabetes, reduced response to insulin, etc.).

Follow all subjects eligible to continue the study and at least 12 participants, 30 days after the first glucose load curve, will be subjected to the second administration of the standard glucose solution according to the procedures described above.

After 15 days, the same subjects will be given a portion of pasta (food on which to measure the glycemic index) containing 50 grams of available carbohydrates. The determination of the quantity of carbohydrates inside the product (pasta) on which it determines the glycemic index must be done with a direct method and supplied by the food company together with the pasta samples. The subject will be invited to consume the pasta in 15 minutes while sipping 200 cc of mineral water at the same time. Blood samples for the determination of blood sugar and insulin will be collected at time 0, and then at 15, 30, 45, 60, 90 and 120 minutes from the start of the pasta intake.

After another 30 days, the third glucose response curve and all insulin will be performed on each subject, with the other modalities of the first two loading curves (this provides an average value of the subject's response to glucose over time).

Phase 3: Statistical processing of the results of phase 2 and determination of the glycemic index and insulinemic index for each type of pasta tested.

Phase 4: For each type of pasta tested, a detailed report will be drawn up, complete with graphs relating to the glycemic and insulinemic response for each subject. Each report will include the glycemic and insulinemic index values of the product concerned.

This will allow to determine which pasta format and which type of flour has the lowest glycemic and insulinemic index.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* No carbohydrate intolerance or diabetes

Exclusion Criteria:

* Intolerance ascertained to the products in study (celiac syndrome)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic Index determination | 1 year
  determination of the glycemic index for the product in study

SECONDARY OUTCOMES:
Insulinemic Index determination | 1 year
  determination of the glycemic index for the product in study

OTHER OUTCOMES:
Best cereal made product identification | 1,5 years
  determination of the pasta format and the type of flour with a lower glycemic and insulinemic index